CLINICAL TRIAL: NCT06663683
Title: Comparative Effects of Hip Thrust Versus Back Squats Resistance Training on Strength, Power and Speed Among Footballer Players
Brief Title: Comparative Effects of Hip Thrust Versus Back Squats Resistance Training Among Footballer Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0428
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Sports Physical Therapy
Keywords: Back Squats; Countermovement Jump; Hip Thrust; Resistance Training; Sprint, Strength

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip thrust (Experimental): The subjects in Hip thrust group will be instructed to perform low-load gluteus activation exercises, which included single-leg bridges, clamshells and quadruped hip extensions. One set of ten repetitions or steps will perform for each exercise. In this training program three stages which focused on enhancing hypertrophy and strength of the hip extensors in sequence. During the training period, the subjects will be instructed to maintain their usual daily activities and diet. All subjects will complete 18 sessions at a frequency of 3 sessions per week and with at least 48 hours between the sessions. Hip thrust training 3 sets with 10 repetitions in each set and 2 minutes rest between each set.
  Interventions: Other: Hip thrust
- Back squat (Experimental): In Back Squat (BS) resistance training the subjects starts with the standing position with the feet flat on the floor, the knees and hips in a neutral, extended anatomical position, and the spine in an upright position with preservation of its natural curves. The squat movement will begin with the descent phase as the hips, knee and ankles flex. A common instruction will be given to the subjectsto descend until the top of the thigh is at least parallel with ground and the hip joint is at least level with or slightly below the knee joint. All subjects will complete 18 sessions at a frequency of 3 sessions per week and with at least 48 hours between sessions. Back squat training 3 sets with 10 repetitions in each set & 2 minutes rest between each set.
  Interventions: Other: Back squat

INTERVENTIONS:
Other: Hip thrust — The subjects in Hip Thrust (HT) group will be instructed to perform low-load gluteus activation exercises, which included single-leg bridges, clamshells and quadruped hip extensions. One set of ten repetitions or steps will perform for each exercise. In this training program three stages which focused on enhancing hypertrophy and strength of the hip extensors in sequence. During the training period, the subjects will be instructed to maintain their usual daily activities and diet. All subjects will complete 18 sessions at a frequency of 3 sessions per week and with at least 48 hours between the sessions. Hip thrust training 3 sets with 10 repetitions in each set and 2 minutes rest between each set.
  Arms: Hip thrust
Other: Back squat — In Back Squat (BS) resistance training the subjects starts with the standing position with the feet flat on the floor, the knees and hips in a neutral, extended anatomical position, and the spine in an upright position with preservation of its natural curves. The squat movement will begin with the descent phase as the hips, knee and ankles flex. A common instruction will be given to the subjects to descend until the top of the thigh is at least parallel with ground and the hip joint is at least level with or slightly below the knee joint. All subjects will complete 18 sessions at a frequency of 3 sessions per week and with at least 48 hours between sessions. Back squat training 3 sets with 10 repetitions in each set & 2 minutes rest between each set.
  Arms: Back squat

SUMMARY:
The purpose of this study is to find which resistance training program hip thrust or back squats will enhance the performance that benefits the strength, power and speed in football players.

DETAILED DESCRIPTION:
In previous study there is less literature in determining the comparative effect of hip thrust and back squat resistance training on performance among footballer players. Therefore there is a dire need to explore the effects of these resistance training exercises. This study aims to observe the effect of hip thrust and back squat resistance training on strength, power and speed in footballer players.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 16-25 years
* Resistance Training of minimum 3 sessions per week
* Experienced players who are in practice from last 1.5 years.

Exclusion Criteria:

* No history of Metabolic Disorders.
* No history of Lower extremity trauma
* Past Surgeries of Spine
* Recreational Players will be excluded

Ages: 16 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Males
Enrollment: 24 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Body Fat Caliper Mass Measurement | 6 weeks
  Body composition measurement is an important assessment technique in sports. Body composition parameters can provide valuable information regarding the amount and ratios of certain tissue components within the body depending on the instrumentation used. In general, parameters such as body fat percentage, fat-free mass, and lean body mass are measured directly, or estimated based on prediction equations or indirect measurements. Skinfold measurement utilizes a caliper to obtain a measure of subcutaneous adiposity (skinfold thickness) at selected sites throughout the body using a double fold of gripped skin
1-Repetition Maximum | 6 weeks
  1-Repetition Maximum is the gold standard for evaluating strength and defined as maximal weight that can be lifted once while maintaining the correct lifting technique. In 1-Repetition maximum eccentric actions are usually coupled with concentric actions which is more reflective of dynamic muscle actions that are commonly used in resistance training and of natural movement in most activities of sports and daily living. This measure has high test-retest reliability of ICC >0.91
Countermovement Jump Test | 6 weeks
  Countermovement Jump Test is commonly used for monitoring status (supercompensation on performance, strength and power muscle) from the analysis of bilateral mechanics and the ability to absorb ground reaction forces by the lower extremity. Conversely, it is expected that the vertical performance is strongly linked to the mechanical variables responsible for the force production, and in turn, the contribution of the elastic elements and joint stability. Intra rater class reliability of countermovement jump test=0.903 to 0.934
Sprint Test | 6 weeks
  Sprint test require skill characteristics that involve the capacity to produce higher velocities to run a set distance within a lower time. Furthermore, this can require the capacity to generate maximal force and power in the direction of running. The profile can be divided into three phases and obtaining their mechanical descriptions can improve the athletes sporting performance and prevent injuries. The aim of this test is to determine quickness of ICC >0.987

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Aftab, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miranda-Oliveira P, Branco M, Fernandes O. Accuracy and Interpretation of the Acceleration from an Inertial Measurement Unit When Applied to the Sprint Performance of Track and Field Athletes. Sensors (Basel). 2023 Feb 4;23(4):1761. doi: 10.3390/s23041761. PMID 36850357
- [Background] Haugen TA, Breitschadel F, Wiig H, Seiler S. Countermovement Jump Height in National-Team Athletes of Various Sports: A Framework for Practitioners and Scientists. Int J Sports Physiol Perform. 2021 Feb 1;16(2):184-189. doi: 10.1123/ijspp.2019-0964. Epub 2020 Nov 20. PMID 33217727
- [Background] Jagim AR, Tinsley GM, Merfeld BR, Ambrosius A, Khurelbaatar C, Dodge C, Carpenter M, Luedke J, Erickson JL, Fields JB, Jones MT. Validation of skinfold equations and alternative methods for the determination of fat-free mass in young athletes. Front Sports Act Living. 2023 Aug 11;5:1240252. doi: 10.3389/fspor.2023.1240252. eCollection 2023. PMID 37637224
- [Background] Gonzalez-Garcia J, Morencos E, Balsalobre-Fernandez C, Cuellar-Rayo A, Romero-Moraleda B. Effects of 7-Week Hip Thrust Versus Back Squat Resistance Training on Performance in Adolescent Female Soccer Players. Sports (Basel). 2019 Apr 3;7(4):80. doi: 10.3390/sports7040080. PMID 30987169
- [Background] Jarosz J, Krolikowska P, Matykiewicz P, Aschenbrenner P, Ewertowska P, Krzysztofik M. Effects of Flywheel vs. Free-Weight Squats and Split Squats on Jumping Performance and Change of Direction Speed in Soccer Players. Sports (Basel). 2023 Jun 23;11(7):124. doi: 10.3390/sports11070124. PMID 37505611
- [Background] Barbalho M, Coswig V, Souza D, Serrao JC, Hebling Campos M, Gentil P. Back Squat vs. Hip Thrust Resistance-training Programs in Well-trained Women. Int J Sports Med. 2020 May;41(5):306-310. doi: 10.1055/a-1082-1126. Epub 2020 Jan 23. PMID 31975359
- [Background] Orjalo AJ, Callaghan SJ, Lockie RG. The Effects of the Barbell Hip Thrust on Post-Activation Performance Enhancement of Change of Direction Speed in College-Aged Men and Women. Sports (Basel). 2020 Nov 24;8(12):151. doi: 10.3390/sports8120151. PMID 33255275
- [Background] Williams MJ, Gibson NV, Sorbie GG, Ugbolue UC, Brouner J, Easton C. Activation of the Gluteus Maximus During Performance of the Back Squat, Split Squat, and Barbell Hip Thrust and the Relationship With Maximal Sprinting. J Strength Cond Res. 2021 Jan 1;35(1):16-24. doi: 10.1519/JSC.0000000000002651. PMID 33332802
- [Background] Plotkin DL, Rodas MA, Vigotsky AD, McIntosh MC, Breeze E, Ubrik R, Robitzsch C, Agyin-Birikorang A, Mattingly ML, Michel JM, Kontos NJ, Lennon S, Fruge AD, Wilburn CM, Weimar WH, Bashir A, Beyers RJ, Henselmans M, Contreras BM, Roberts MD. Hip thrust and back squat training elicit similar gluteus muscle hypertrophy and transfer similarly to the deadlift. Front Physiol. 2023 Oct 9;14:1279170. doi: 10.3389/fphys.2023.1279170. eCollection 2023. PMID 37877099
- [Background] Oliver JL, Ramachandran AK, Singh U, Ramirez-Campillo R, Lloyd RS. The Effects of Strength, Plyometric and Combined Training on Strength, Power and Speed Characteristics in High-Level, Highly Trained Male Youth Soccer Players: A Systematic Review and Meta-Analysis. Sports Med. 2024 Mar;54(3):623-643. doi: 10.1007/s40279-023-01944-8. Epub 2023 Oct 28. PMID 37897637
- [Background] Querido SM, Clemente FM. Analyzing the effects of combined small-sided games and strength and power training on the fitness status of under-19 elite football players. J Sports Med Phys Fitness. 2020 Jan;60(1):1-10. doi: 10.23736/S0022-4707.19.09818-9. PMID 32008309
- [Background] Hammond A, Perrin C, Steele J, Giessing J, Gentil P, Fisher JP. The effects of a 4-week mesocycle of barbell back squat or barbell hip thrust strength training upon isolated lumbar extension strength. PeerJ. 2019 Jul 26;7:e7337. doi: 10.7717/peerj.7337. eCollection 2019. PMID 31388473
- [Background] Millar NA, Colenso-Semple LM, Lockie RG, Marttinen RHJ, Galpin AJ. In-Season Hip Thrust vs. Back Squat Training in Female High School Soccer Players. Int J Exerc Sci. 2020 Feb 1;13(4):49-61. doi: 10.70252/UELS8581. eCollection 2020. PMID 32148631
- [Background] Otsuka M, Honjo T, Nagano A, Isaka T. Kinetics in lumbosacral and lower-limb joints of sprinters during barbell hip thrust compared to deadlift and back squat. PLoS One. 2021 Jul 1;16(7):e0251418. doi: 10.1371/journal.pone.0251418. eCollection 2021. PMID 34197487